CLINICAL TRIAL: NCT00689988
Title: Augmentative and Alternative Communication and Lexical Gain in Children With Down Syndrome: Pilot Study
Brief Title: Augmentative and Alternative Communication (AAC) and Lexical Gain in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Suelly Cecilia Olivan Limongi, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05/1149
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Down Syndrome
Keywords: Down syndrome; communication AIDS for disabled; language development disorders; vocabulary; gestures; language tests; child
MeSH Terms: conditions — Down Syndrome; Language Development Disorders; Gestures | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SG (Experimental): Study Group: five children with Down syndrome submitted to speech-language intervention with AAC intervention
  Interventions: Behavioral: speech-language therapy with AAC intervention

INTERVENTIONS:
Behavioral: speech-language therapy with AAC intervention — speech-language intervention in weekly 40-minutes sessions, without the presence of parents or caregivers, and 5 to 10-minutes to parents training and orientation

SUMMARY:
Children with Down syndrome (DS) have language development particularities that have negative effects in the communication capacity. By this way, Augmentative and Alternative Communication (AAC) is indicated to this population. The aim of this study was to verify the AAC impact in the lexical gain of children with DS.

DETAILED DESCRIPTION:
Five children with DS, with the same cognitive level, participated in this study. Longitudinal follow-up of twelve months of speech-language therapy with AAC use was undertaken. A lexical evaluation was done at the beginning and the end of this follow-up. Correct responses in the lexical evaluation were increased, but not necessarily in the spoken modality. The comparisons showed significant results in use of substitutions processes, and to no-answers.

ELIGIBILITY:
Inclusion Criteria:

* genetic diagnosis of Down syndrome
* be at the preoperational period
* good health conditions
* expressive language impairment (communication by vocal and gestures, predominantly)

Exclusion Criteria:

* presence of major malformations
* presence of another genetic syndrome
* severe neonatal asphyxia, hearing impairment or visual

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2005-07; Primary Completion 2007-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Performance on a initial and final lexical assessments, after 12 months of speech-language therapy | 12 months

SECONDARY OUTCOMES:
Performance on longitudinal follow-up of twelve months of speech-language therapy with AAC use | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra CF Pires, PhD student, Principal Investigator — University of Sao Paulo; Suelly CO Limongi, PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo - School of Medicine - Department of Physiotherapy, Communication Sciences and Disorders, Occupational Therapy, São Paulo, São Paulo, Brazil